CLINICAL TRIAL: NCT03233412
Title: Ensaio clínico Randomizado Avaliando a eficácia do Tratamento tópico Com Imiquimode em lesões Intraepiteliais Cervicais de Alto Grau
Brief Title: Randomized Clinical Trial Evaluating the Efficacy of Topical Imiquimod in High Grade Cervical Intraepithelial Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BarretosCH-20171
Record Dates: First submitted 2017-07-06; First posted 2017-07-28 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2019-04

CONDITIONS: High Grade Intraepithelial Neoplasia; Cervix Cancer
Keywords: high grade cervical intraepithelial neoplasia; Immunomodulatory treatment
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Imiquimod

STUDY DESIGN:
Intervention Model Description: Patients between 25 and 50 years old with histological diagnosis of high-grade intraepithelial lesion, obtained through satisfactory colposcopy and without previous treatment, who will be selected in the preventive clinic of the Hospital de Cancer de Barretos-SP (HCB ). Eligible patients will be identified at the return visit, when they will come to the hospital to check the result of the examination. In this study the patients will be randomized into two groups: Group 1: Control, where standard treatment will be offered, which is the conization of the uterine cervix with loop electrosurgical excision procedure(LEEP); Group 2: experimental group, which will receive topical treatment in the uterine cervix with immunomodulator (Imiquimod), for a period of 12 weeks, with weekly applications (1x / week). 30 to 60 days after immunomodulatory treatment the patient will be submitted to standard treatment with cervical conization with LEEP.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Will be offered the standard treatment, which is the conization of the uterine cervix with loop electrosurgical excision procedure (LEEP).
  Interventions: Procedure: Control
- Imiquimod (Experimental): Will receive topical uterine cervix (Imiquimod) treatment for a period of 12 weeks with weekly applications (1x / week). 30-60 days afterwards they will be submitted to standard treatment with conization of the uterine cervix with loop electrosurgical excision procedure (LEEP).
  Interventions: Procedure: Control; Drug: Imiquimod

INTERVENTIONS:
Procedure: Control — Exertion of the cervix transformation zone
  Other Names: loop electrosurgical excision procedure; Conization of the cervix
Drug: Imiquimod — Application by the doctor of immunomodulatory cream on the uterine cervix 1 time per week for 12 weeks
  Other Names: Imiquimod 5% cream; Ixium 5%
  Arms: Imiquimod

SUMMARY:
Cervical cancer is one of the leading malignancies affecting women, with 311,000 deaths in 2018, most of them seen in underdeveloped countries. This neoplasm has a pre-invasive state, such as cervical intraepithelial neoplasia (CIN), which is caused by HPV (Human Papillomavirus) infection. The female organism most often is able to eliminate the virus, especially in young patients. However, when the infection becomes persistent, especially for subtypes 16 and 18, the risk of CIN developing an increased. Cytological screening programs can efficiently and wirelessly do this. As high-grade intraepithelial lesions (CIN 2/3) are as demonstrated by worse regression rate, only 13.3% at one year, and higher risk for progression to invasive cancer. As CIN 2/3 need treatment, and as more therapies as they are excisional, which theoretically are better, however, they may compromise the reproductive future of women who are unthreatened, increasing the risk of preterm labor, premature rupture of amniotic membranes, low weight Birth and perinatal mortality. This relationship aroused interest in seeking alternative therapies. Decrease antiviral activity directed against HPV, associated with a higher rate of elimination of the infection. Immediate, an agent that stimulates like dendritic cells to producer cytokines and activates epithelial T cells. Imiquimode, when used in vulvar neoplasias, has been shown to be effective, presenting satisfactory results without treatment of CIN 2/3 of the uterine cervix, requiring a better scientific compilation. Based on these data, this study aims to evaluate the efficacy of topical immunomodulatory treatment for high-grade cervical intraepithelial lesions.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 25 and 50 with histological diagnosis of CIN 2/3;
* Living 300 km or less from the city of Barretos-São Paulo / Brazil.

Exclusion Criteria:

* Suspected adenocarcinoma (in situ or invasive) or invading squamous cell carcinoma by colposcopy and/or citology;
* Being pregnant or breastfeeding;
* Women with some immunodeficiency or transplanted;
* Previous treatment history for CIN 2/3.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of immunomodulatory treatment with Imiquimod in high grade intraepithelial lesions of the cervix compared to standard electrosurgical excision procedure (LEEP) treatment. | 30 months
  We will evaluate the efficacy of the Imiquimod treatment applied by the physician after histological examination of the uterine cervix obtained by electrosurgical excision procedure (LEEP) and compare the rate of relapse / reoperation with the control patient only submitted to the standard treatment with LEEP

SECONDARY OUTCOMES:
Local and systemic adverse events | 30 months
  To assess the local and systemic adverse effects of topical immunomodulatory treatment through anamnesis and physical examination.
Compare CIN 2 and CIN 3 for the difference in response to immunomodulatory treatment | 30 months
  It will be evaluated separately from the results of the treatment response with Imiquimod in CIN 2 and CIN 3 lesions.
Definition of the difference in cost from actual standard treatment compared to Imiquimod | 30 months
  The value in Brazilian reais of treatment with Imiquimod will be defined as compared to the amount spent for the standard treatment with LEEP
Evaluation of recurrence of high grade cervical squamous intraepithelial lesion after 2 years of treatment. | 24 months
  To evaluate the recurrence after 2 years of the end of the immunomodulatory topical treatment.
Evaluation of reoperation rate after immunomodulatory treatment associated with standard treatment with LEEP compared to LEEP alone. | 24 months
  Evaluation of reoperation rate in post-treatment follow-up.
Clearance HPV | 30 months
  To evaluate the persistence or not of the HPV virus and which specific type to relate to the efficacy of the immunomodulatory treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D Reis, PhD, Study Director — Barretos Cancer Hospital; Bruno DO Fonseca, MD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American College of Obstetricians and Gynecologists. Practice Bulletin No. 140: management of abnormal cervical cancer screening test results and cervical cancer precursors. Obstet Gynecol. 2013 Dec;122(6):1338-67. doi: 10.1097/01.AOG.0000438960.31355.9e. No abstract available. PMID 24264713
- [Result] Martin-Hirsch PP, Paraskevaidis E, Bryant A, Dickinson HO, Keep SL. Surgery for cervical intraepithelial neoplasia. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD001318. doi: 10.1002/14651858.CD001318.pub2. PMID 20556751
- [Result] Lin CT, Qiu JT, Wang CJ, Chang SD, Tang YH, Wu PJ, Jung SM, Huang CC, Chou HH, Jao MS, Lai CH. Topical imiquimod treatment for human papillomavirus infection in patients with and without cervical/vaginal intraepithelial neoplasia. Taiwan J Obstet Gynecol. 2012 Dec;51(4):533-8. doi: 10.1016/j.tjog.2012.09.006. PMID 23276555
- [Result] Pachman DR, Barton DL, Clayton AC, McGovern RM, Jefferies JA, Novotny PJ, Sloan JA, Loprinzi CL, Gostout BS. Randomized clinical trial of imiquimod: an adjunct to treating cervical dysplasia. Am J Obstet Gynecol. 2012 Jan;206(1):42.e1-7. doi: 10.1016/j.ajog.2011.06.105. Epub 2011 Jul 13. PMID 21907959
- [Result] McCredie MR, Sharples KJ, Paul C, Baranyai J, Medley G, Jones RW, Skegg DC. Natural history of cervical neoplasia and risk of invasive cancer in women with cervical intraepithelial neoplasia 3: a retrospective cohort study. Lancet Oncol. 2008 May;9(5):425-34. doi: 10.1016/S1470-2045(08)70103-7. Epub 2008 Apr 11. PMID 18407790
- [Result] Arbyn M, Kyrgiou M, Simoens C, Raifu AO, Koliopoulos G, Martin-Hirsch P, Prendiville W, Paraskevaidis E. Perinatal mortality and other severe adverse pregnancy outcomes associated with treatment of cervical intraepithelial neoplasia: meta-analysis. BMJ. 2008 Sep 18;337:a1284. doi: 10.1136/bmj.a1284. PMID 18801868
- [Result] Kyrgiou M, Koliopoulos G, Martin-Hirsch P, Arbyn M, Prendiville W, Paraskevaidis E. Obstetric outcomes after conservative treatment for intraepithelial or early invasive cervical lesions: systematic review and meta-analysis. Lancet. 2006 Feb 11;367(9509):489-98. doi: 10.1016/S0140-6736(06)68181-6. PMID 16473126
- [Result] Jin G, LanLan Z, Li C, Dan Z. Pregnancy outcome following loop electrosurgical excision procedure (LEEP) a systematic review and meta-analysis. Arch Gynecol Obstet. 2014 Jan;289(1):85-99. doi: 10.1007/s00404-013-2955-0. Epub 2013 Jul 11. PMID 23843155
- [Result] Insinga RP, Dasbach EJ, Elbasha EH. Epidemiologic natural history and clinical management of Human Papillomavirus (HPV) Disease: a critical and systematic review of the literature in the development of an HPV dynamic transmission model. BMC Infect Dis. 2009 Jul 29;9:119. doi: 10.1186/1471-2334-9-119. PMID 19640281
- [Result] Kocken M, Helmerhorst TJ, Berkhof J, Louwers JA, Nobbenhuis MA, Bais AG, Hogewoning CJ, Zaal A, Verheijen RH, Snijders PJ, Meijer CJ. Risk of recurrent high-grade cervical intraepithelial neoplasia after successful treatment: a long-term multi-cohort study. Lancet Oncol. 2011 May;12(5):441-50. doi: 10.1016/S1470-2045(11)70078-X. PMID 21530398
- [Result] Conner SN, Cahill AG, Tuuli MG, Stamilio DM, Odibo AO, Roehl KA, Macones GA. Interval from loop electrosurgical excision procedure to pregnancy and pregnancy outcomes. Obstet Gynecol. 2013 Dec;122(6):1154-9. doi: 10.1097/01.AOG.0000435454.31850.79. PMID 24201682
- [Result] Spracklen CN, Harland KK, Stegmann BJ, Saftlas AF. Cervical surgery for cervical intraepithelial neoplasia and prolonged time to conception of a live birth: a case-control study. BJOG. 2013 Jul;120(8):960-5. doi: 10.1111/1471-0528.12209. Epub 2013 Mar 14. PMID 23489374
- [Result] Grimm C, Polterauer S, Natter C, Rahhal J, Hefler L, Tempfer CB, Heinze G, Stary G, Reinthaller A, Speiser P. Treatment of cervical intraepithelial neoplasia with topical imiquimod: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):152-9. doi: 10.1097/AOG.0b013e31825bc6e8. PMID 22914404
- [Result] Mathiesen O, Buus SK, Cramers M. Topical imiquimod can reverse vulvar intraepithelial neoplasia: a randomised, double-blinded study. Gynecol Oncol. 2007 Nov;107(2):219-22. doi: 10.1016/j.ygyno.2007.06.003. Epub 2007 Jul 25. PMID 17655918
- [Result] van Seters M, van Beurden M, ten Kate FJ, Beckmann I, Ewing PC, Eijkemans MJ, Kagie MJ, Meijer CJ, Aaronson NK, Kleinjan A, Heijmans-Antonissen C, Zijlstra FJ, Burger MP, Helmerhorst TJ. Treatment of vulvar intraepithelial neoplasia with topical imiquimod. N Engl J Med. 2008 Apr 3;358(14):1465-73. doi: 10.1056/NEJMoa072685. PMID 18385498
- [Result] van Seters M, van Beurden M, de Craen AJ. Is the assumed natural history of vulvar intraepithelial neoplasia III based on enough evidence? A systematic review of 3322 published patients. Gynecol Oncol. 2005 May;97(2):645-51. doi: 10.1016/j.ygyno.2005.02.012. PMID 15863172
- [Result] Chen FP. Efficacy of imiquimod 5% cream for persistent human papillomavirus in genital intraepithelial neoplasm. Taiwan J Obstet Gynecol. 2013 Dec;52(4):475-8. doi: 10.1016/j.tjog.2013.10.004. PMID 24411029
- [Result] Diaz-Arrastia C, Arany I, Robazetti SC, Dinh TV, Gatalica Z, Tyring SK, Hannigan E. Clinical and molecular responses in high-grade intraepithelial neoplasia treated with topical imiquimod 5%. Clin Cancer Res. 2001 Oct;7(10):3031-3. PMID 11595691
- [Result] Gunderson CC, Nugent EK, Elfrink SH, Gold MA, Moore KN. A contemporary analysis of epidemiology and management of vaginal intraepithelial neoplasia. Am J Obstet Gynecol. 2013 May;208(5):410.e1-6. doi: 10.1016/j.ajog.2013.01.047. Epub 2013 Feb 1. PMID 23380265
- [Result] Haidopoulos D, Diakomanolis E, Rodolakis A, Voulgaris Z, Vlachos G, Intsaklis A. Can local application of imiquimod cream be an alternative mode of therapy for patients with high-grade intraepithelial lesions of the vagina? Int J Gynecol Cancer. 2005 Sep-Oct;15(5):898-902. doi: 10.1111/j.1525-1438.2005.00152.x. PMID 16174242
- [Result] Darragh TM, Colgan TJ, Cox JT, Heller DS, Henry MR, Luff RD, McCalmont T, Nayar R, Palefsky JM, Stoler MH, Wilkinson EJ, Zaino RJ, Wilbur DC; Members of LAST Project Work Groups. The Lower Anogenital Squamous Terminology Standardization Project for HPV-Associated Lesions: background and consensus recommendations from the College of American Pathologists and the American Society for Colposcopy and Cervical Pathology. Arch Pathol Lab Med. 2012 Oct;136(10):1266-97. doi: 10.5858/arpa.LGT200570. Epub 2012 Jun 28. PMID 22742517
- [Result] International Agency for Research on Cancer, World Health Organization, Globocan, Estimated Cancer Incidence, Mortality and Prevalence Worldwide in 2012
- [Derived] Fonseca BO, Possati-Resende JC, Salcedo MP, Schmeler KM, Accorsi GS, Fregnani JHTG, Antoniazzi M, Pantano NP, Santana IVV, Matsushita GM, Dos Reis R. Topical Imiquimod for the Treatment of High-Grade Squamous Intraepithelial Lesions of the Cervix: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):1043-1053. doi: 10.1097/AOG.0000000000004384. PMID 33957649